CLINICAL TRIAL: NCT01746849
Title: Phase II Study of Palifermin With Leuprolide Acetate or Degarelix For the Promotion of Immune Recovery Following Total Body Irradiation Based T-Cell Depleted Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Palifermin With Leuprolide Acetate for the Promotion of Immune Recovery Following Total Body Irradiation Based T-Cell Depleted Allogeneic Hematopoietic Stem Cell Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-077
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Leukemia; Multiple Myeloma; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma
Keywords: LUPRON DEPOT; PALIFERMIN; 12-077
MeSH Terms: conditions — Leukemia; Multiple Myeloma; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin | interventions — Fibroblast Growth Factor 7; Leuprolide; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation; Thiotepa; Cyclophosphamide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

ARMS (2):
- palifermin with Lupron (Experimental): All patients undergo total body irradiation (TBI) on days -9 to -6 & receive thiotepa intravenously (IV) over 2-4 hours on days -5 to -4, cyclophosphamide IV over 30-60 minutes on days -3 to -2, & anti-thymocyte globulin infused over 12 hours on days -3 to -2 Pts undergo T-cell depleted allogeneic hematopoietic stem cell transplant on day 0. Pts will receive a three month depot dose of Lupron 3-6 weeks prior to the start date of the pre-transplant conditioning regimen. Pts will receive palifermin at 60mcg/kg/day IV on three consecutive days, 24 hours apart with the last dose administered no less than 24 & no more than 48 hours prior to the start of cytoreduction. Pts will receive three additional daily doses of palifermin the first approximately 6 hours after the stem cell infusion on day 0, followed by two daily doses given at 24 hour intervals on d+1 & d+2. Pts will receive a further 3-month depot injection of Lupron approximately 3 months (+/- one week) post the first dose.
  Interventions: Biological: Palifermin; Biological: Lupron; Procedure: peripheral blood stem cell transplantation; Radiation: Total-Body Irradiation (TBI); Drug: Thiotepa; Drug: Cyclophosphamide
- palifermin with Degarelix (Experimental): Participants on the degarelix arm will receive a loading dose of degarelix 240 mcg subcutaneous 4-14 days before the start of pre-transplant conditioning. All participants will receive palifermin at 60mcg/kg/day IV on three consecutive days, 24 hours apart with the last dose administered no less than 24 and no more than 48 hours prior to the start of cytoreduction.
  Interventions: Biological: Palifermin; Procedure: peripheral blood stem cell transplantation; Radiation: Total-Body Irradiation (TBI); Drug: Thiotepa; Drug: Cyclophosphamide; Drug: Degarelix

INTERVENTIONS:
Biological: Palifermin
Biological: Lupron
  Arms: palifermin with Lupron
Procedure: peripheral blood stem cell transplantation
Radiation: Total-Body Irradiation (TBI)
Drug: Thiotepa
Drug: Cyclophosphamide
Drug: Degarelix
  Arms: palifermin with Degarelix

SUMMARY:
The purpose of this study is to help determine if palifermin and leuprolide acetate can help the immune system recover faster following a stem cell transplant. Blood stem cells are very young blood cells that grow in the body to become red or white blood cells or platelets. The transplant uses stem cells in the blood from another person. The donor can be a family member or a volunteer donor. This is called an allogeneic stem cell transplant.

The investigators want to see if palifermin and leuprolide acetate can help the immune system recover faster after an allogenic transplant because experiments have shown they may be able to do this.

DETAILED DESCRIPTION:
Patients will be randomized to one of two arms: palifermin with Lupron, and control. The control arm consists of a standard TCD allo-HSCT without the addition of palifermin or Lupron.

Patients randomized to receive Lupron will receive a three month depot dose 3-6 weeks prior to the start date of the pre-transplant conditioning regimen. Patients assigned to receive palifermin will receive this drug at 60mcg/kg/day IV on three consecutive days, 24 hours apart with the last dose administered no less than 24 and no more than 48 hours prior to the start of cytoreduction. The preparative regimen to be used for transplants will consist of: hyperfractionated TBI administered in 11 doses over 4 days for a total of 1375 cGy, thiotepa 5 mg/kg/day IV x 2 days and cyclophosphamide with mesna prophylaxis 60 mg/kg/day IV x 2 days. All patients will receive ATG for two doses prior to transplant, except recipients of mismatched grafts (in the GVHD vector) will receive three doses. G-CSF mobilized CD34 PBSCs obtained from the HLA compatible donor will be infused on day 0. Patients assigned to receive palifermin will receive three additional daily doses of the drug, the first approximately 6 hours after the stem cell infusion on day 0, followed by two daily doses given at 24 hour intervals on d+1 and d+2. Patients assigned to receive Lupron will receive a further 3-month depot injection approximately 3 months (+/- one week) post the first dose. Supportive care will be administered as per the BMT Service guidelines. The conditioning regimen may be modified to allow an extra day during conditioning or prior to the graft infusion if required by donor and/or patient scheduling restrictions.

ELIGIBILITY:
Inclusion Criteria:

Treatment Portion:

* AML in 1st remission - for patients whose AML does not have "good risk" cytogenetic features (i.e. t (8;21), t(15;17), inv 16 without c-kit mutations).
* Acute leukemias of ambiguous lineage in ≥ 1st remission
* Secondary AML in remission
* AML in ≥ 2nd remission
* ALL in 1st remission with clinical or molecular features indicating a high risk for relapse; or ALL ≥ 2nd remission
* CML failing to respond to or not tolerating imatinib, dasatinib or nilotinib in first chronic phase of disease; CML in accelerated phase, second chronic phase, or in CR after accelerated phase or blast crisis.
* Non-Hodgkins lymphoma with chemo responsive disease in any of the following categories:

intermediate or high grade lymphomas who have failed to achieve a first CR or have relapsed following a 1st remission who are not candidates for autologous transplants.

b.ii. any NHL in remission which is considered not curable with chemotherapy alone and not eligible/appropriate for autologous transplant.

* Myelodysplastic syndrome (MDS): RA/RCMD with high risk cytogenetic features or transfusion dependence, RAEB-1 and RAEB-2
* Chronic myelomonocytic leukemia: CMML-1 and CMML-2.
* Patient's age is ≥18 or ≤60 years old
* Patients must have a Karnofsky (adult) or Lansky (pediatric) Performance Status ≥ 70%
* Patients must have adequate organ function measured by:

Cardiac: asymptomatic or if symptomatic then LVEF at rest must be > 50% and must improve with exercise.

* Pulmonary: asymptomatic or if symptomatic, DLCO > 60% of predicted (corrected for hemoglobin)
* Hepatic: < 3xULN ALT and < 1.5 total serum bilirubin, unless there is congenital benign hyperbilirubinemia
* Renal: serum creatinine < 1.2 mg/dL or if serum creatinine is outside the normal range, the CrCl > 50 ml/min (measured or calculated/estimated)
* Patients have a plan to receive a CD34-selected peripheral blood stem cell transplant with TBI-based conditioning.

Exclusion Criteria:

* Active extramedullary disease
* Active and uncontrolled infection at time of transplantation
* Patients who have undergone a prior allogeneic or autologous stem cell transplant within the previous six months.
* Pregnant or breast feeding
* HIV infection
* Patient is felt to not be a candidate for TBI by the BMT service

Donor Inclusion Criteria:

* Donor must be willing and able to undergo PBSC collection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2012-12; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
a CD4+ T cell count of greater than 200 | 6 months
  Will be documented by flow cytometry performed in the clinical lab on peripheral blood.

SECONDARY OUTCOMES:
Overall Survival | 2 years
  Overall survival is defined as the time from transplant to death of last follow-up.
Transplant Related Mortality | 6 months
  TRM is defined as death at any time from the commencement of pre-transplant conditioning due to any cause other than disease relapse with the exception of automobile or other accidents.
Incidence of infections | 2 years
  Any bacterial, viral, fungal or parasitic infection that necessitates therapy will be noted.
Relapse | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Perales, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/